CLINICAL TRIAL: NCT00013052
Title: Improving Health Outcomes of Diabetic Veterans: A Diabetic Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: DII 99-097
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Peer led classes. Led by trained veterans with a chronic disease.

INTERVENTIONS:
Behavioral: Peer led classes. Led by trained veterans with a chronic disease.

SUMMARY:
Control of the blood sugar prevents complications and results in extra years of life in patients with diabetes. Practice Guidelines delineating specific ways physicians manage diabetes have been outlined. Missing are guidelines for health care providers to encourage patients to take responsibility for their diabetes. Traditional patient education models have been ineffective in managing diabetic persons because they have relied upon information given alone and are disease centered rather than patient centered. This study will explore the role of self-efficacy in helping veterans move toward healthy behaviors.

DETAILED DESCRIPTION:
Background:

Control of the blood sugar prevents complications and results in extra years of life in patients with diabetes. Practice Guidelines delineating specific ways physicians manage diabetes have been outlined. Missing are guidelines for health care providers to encourage patients to take responsibility for their diabetes. Traditional patient education models have been ineffective in managing diabetic persons because they have relied upon information given alone and are disease centered rather than patient centered. This study will explore the role of self-efficacy in helping veterans move toward healthy behaviors.

Objectives:

The long-term objectives are to: 1) increase recognition of veteran�s responsibility for health; 2) develop more effective skills in managing chronic conditions; and 3) explore the role of self-efficacy in facilitating improvements in health behaviors and health care utilization.

Methods:

This is a prospective, randomized controlled clinical trial of 2,068 cognitively intact, diabetic veterans. The outcome measures (health behaviors, self-efficacy, health status and health care utilization) will be measured using self-rated scales developed and tested by Lorig and colleagues from Stanford University. Glucose levels and BMI changes will be evaluated using information documented in the medical record.

Status:

Enrollment (a total of 326 patients) is closed. All necessary data have been received and are being analyzed.

ELIGIBILITY:
Inclusion Criteria:

Cognitively intact diabetic veterans.

Exclusion Criteria:

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2068 (Estimated)
Dates: Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Nodhturft, EdD RN, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL; Carolee A. DeVito, PhD MPH, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (3):
- United States (3):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - West Palm Beach VA Medical Center, West Palm Beach, FL, West Palm Beach, Florida

REFERENCES:
- [Result] Nodhturft V, Schneider JM, Hebert P, Bradham DD, Bryant M, Phillips M, Russo K, Goettelman D, Aldahondo A, Clark V, Wagener S. Chronic disease self-management: improving health outcomes. Nurs Clin North Am. 2000 Jun;35(2):507-18. PMID 10873263